CLINICAL TRIAL: NCT06654453
Title: The Thrombus Aspiration During Percutaneous Coronary Intervention After Thrombolysis in ST-elevation Myocardial Infarction
Brief Title: The Thrombus Aspiration During PCI After Thrombolysis in STEMI
Acronym: Optimal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenghua Zhou (Other)
Responsible Party: Sponsor-Investigator, Shenghua Zhou, Director, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYZ20240204
Record Dates: First submitted 2024-10-20; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Thrombus aspiration; Percutaneous coronary intervention; High thrombus burden; Randomized controlled trial
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Thrombectomy; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thrombectomy + PCI Arm (Experimental): This group will receive thrombectomy combined with percutaneous coronary intervention.
  Interventions: Procedure: Thrombectomy; Procedure: Percutaneous Coronary Intervention
- PCI-only Arm (Active Comparator): PCI is an established treatment for STEMI, and you are comparing it to the experimental group that receives an additional thrombectomy procedure.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Thrombectomy — Manual thrombectomy followed by Percutaneous Coronary Intervention (PCI), a procedure involving mechanical removal of thrombus before stent placement in coronary arteries to restore blood flow in STEM
  Arms: Thrombectomy + PCI Arm
Procedure: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention, involving balloon angioplasty and stent placement to open blocked coronary arteries in STEMI patients after thrombolysis.

SUMMARY:
The goal of this clinical trial is to determine whether thrombus aspiration combined with percutaneous coronary intervention (PCI) improves clinical outcomes in ST-segment elevation myocardial infarction (STEMI) patients with high thrombus burden post-thrombolysis, compared to PCI alone. The study population includes 3500 STEMI patients, confirmed by diagnosis, who are transferred to PCI centers after receiving thrombolysis and have no contraindications to thrombolysis.The main questions it aims to answer are:

1. Does thrombus aspiration reduce 30-day major adverse cardiovascular events (MACE), including cardiovascular death, recurrent myocardial infarction, stroke, or heart failure rehospitalization?
2. Can thrombus aspiration improve microcirculation and clinical outcomes for high thrombus burden patients after thrombolysis? Researchers will compare patients randomly assigned to receive thrombus aspiration combined with PCI versus those who receive PCI alone to evaluate the effects on reducing MACE and improving clinical recovery.

Participants will:

Undergo initial thrombolysis followed by transfer to PCI centers. Be randomly assigned in a 1:1 ratio to receive either thrombus aspiration combined with PCI or PCI alone.

Be followed for 30 days post-treatment to assess MACE and other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with STEMI.
2. No contraindications for thrombolysis and has received thrombolytic treatment.
3. Undergoing coronary angiography within 2 to 24 hours post-thrombolysis.
4. Angiographic results confirm TIMI thrombus load ≥ 4 and residual stenosis > 50%.

Exclusion Criteria:

1. Contraindications for thrombolysis.
2. Cardiogenic shock.
3. Need for coronary artery bypass grafting.
4. Age less than 18 years.
5. Life expectancy of less than 6 months.
6. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
30-day Major Adverse Cardiovascular Events (MACE) | From enrollment to the end of treatment at 4 weeks
  A composite of cardiovascular death, recurrent myocardial infarction, stroke, and rehospitalization for heart failure within 30 days post-intervention.

SECONDARY OUTCOMES:
Reperfusion Success | Within 30 minutes post-PCI (Percutaneous Coronary Intervention)
  The percentage of patients achieving successful reperfusion as indicated by TIMI flow grade improvement (e.g., achieving TIMI 2 or 3 flow) after the intervention.
Follow-up MACE at 6 Months | From enrollment to the end of treatment at 6 months
  The rate of major adverse cardiovascular events (including cardiovascular death, myocardial infarction, and stroke) occurring within 6 months post-intervention.
Follow-up all-cause mortality at 6 Months | From enrollment to the end of treatment at 6 months
  The rate of all-cause mortality occurring within 6 months post-intervention.
Follow-up MACE at 12 Months | From enrollment to the end of treatment at 12 months
  The rate of major adverse cardiovascular events (including cardiovascular death, myocardial infarction, and stroke) occurring within 12 months post-intervention.
Follow-up all-cause mortality at 12 Months | From enrollment to the end of treatment at 12 months
  The rate of all-cause mortality occurring within 12 months post-intervention.

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: To access the IPD and supporting information, interested parties should contact the principal investigator or designated study coordinator.